CLINICAL TRIAL: NCT06618807
Title: A Pilot Study Evaluating the Feasibility, Safety, and Efficacy of the Neuro RX Gamma (Version 2) for the Treatment of Mild Cognitive Impairment (MCI)
Brief Title: Infrared Light for Memory Loss in Mild Cognitive Impairment (MCI)
Acronym: PBMCI-Prime
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Corinne Fischer, staff psychiatrist, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB #24-188
Record Dates: First submitted 2024-09-16; First posted 2024-10-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Mild Cognitive Impairment (MCI) Due to Alzheimer's Disease
Keywords: photobiomodulation; light therapy; Alzheimer's Disease; clinical trial; Mild Cognitive Impairment (MCI); home-based treatment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The trial is a randomized, double-blind, sham-controlled trial designed to evaluate the efficacy of transcranial photobiomodulation (tPBM) in improving cognitive function among patients with MCI. Participants will be randomly assigned in a 1:1 ratio to receive either active tPBM treatment or a sham treatment. The trial will evaluate the effects of home-based tPBM sessions daily 6 days/week over 8 weeks on mitochondrial function via Blood-based and Neuroimaging biomarkers in patients with MCI.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To ensure balanced allocation across trial groups, the trial will employ a block randomization method with a block size of 4. This method generates balanced combinations (TTCC, TCTC, TCCT, CTTC, CTCT, CCTT), from which blocks will be randomly selected to assign the 60 participants evenly, with 30 participants per group. Randomization will be performed using a computer-generated process, and an independent Research Assistant will manage this to maintain blinding for participants, study investigators, and data analysts. Unblinding will occur only in the case of patient emergencies or at the end of the trial. This approach ensures that each participant is assigned to either the sham or active treatment group in a 1:1 ratio, while maintaining the integrity of the trial and reducing potential biases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Active Comparator): The active group will undergo a 8-week trial of home-use tPBM using the active Neuro RX Gamma (v2) device, 6 days/week, 20 minutes per session.
  Interventions: Device: Active tPBM device
- Sham group (Sham Comparator): The sham group will undergo a 8-week trial of home-use PBM using the sham Neuro RX Gamma (v2) device, 6 days/week, 20 minutes per session.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: Active tPBM device — The Neuro RX Gamma (version 2) delivers a synchronized pulse frequency of 40 Hz from all LED clusters. The gamma pulse frequency of 40 Hz has been demonstrated to attenuate amyloid beta proteins production in the hippocampus and modulate microglial activity resulting in increased scavenging of amyloid beta which may lead to improving cognition in MCI. Finally, the Vielight Neuro RX Gamma (version 2) has been designed to target the delivery of NIR energy to particular brain regions; specifically the default mode network (DMN). The active intervention device proceeds to deliver light to each LED at 40 Hz with a 50% duty cycle for 20 minutes and stops automatically. During the 20 minute treatment the power indicator LED on the controller flashes green at 40 Hz. The operator is notified that the treatment is finished when the power indicator LED on the controller stops flashing and the device beeps 2 times.
  Arms: Active group
Device: Sham device — The sham device delivers infrared light for only a few seconds before stopping. The controller will still show a green light to maintain the study's blinding. If the headset is removed, the device will emit a beep and cease functioning.
  Arms: Sham group

SUMMARY:
Mild cognitive impairment (MCI) is a transitional risk state that occurs between the normal aging process and Alzheimer's dementia (AD). On average 32% of patients with MCI will progress to dementia, 62% will stay stable, and about 6% will return to normal cognition at subsequent visits.

Current treatment for MCI includes cholinesterase inhibitors (donepezil, galantamine and rivastigmine), and NMDA receptor antagonists (memantine) which delay or slow the worsening of symptoms and treat cognitive symptoms (memory loss, confusion, and problems with thinking and reasoning). Despite currently ongoing drug studies and modest clinical benefits of currently approved drug treatments, there continues to remain a need for treatments for long term symptomatic improvement of MCI with fewer and less severe side effects.

Photobiomodulation (PBM) therapy also called low-level laser (or light) therapy (LLLT) is a safe, non-invasive, non-thermal (no significant heat is generated) method of therapy which uses either visible red or near-infrared (NIR) light to stimulate, heal and repair damaged or dying tissue cells. This study proposes to use the Neuro RX Gamma device (version 2) to deliver NIR light energy to particular brain regions which are dysfunctional in MCI participants.

DETAILED DESCRIPTION:
This study will recruit approximately 60 participants with MCI for the study, and the total expected duration of the participant's participation in the study is 12 weeks. The active and sham Neuro RX gamma device (v2) consists of a headset with a built-in controller and nasal applicator. The nasal applicator contains a single LED and will be placed into the nostril and clipped into place. The headset is a wearable applicator that may be adjusted. It consists of 5 LEDs. A red star symbol identifies the front of the headset and helps the user orientate the headset on the head. LEDs are semiconductor electronic components that emit light.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet the criteria for MCI of 1) cognitive concern by the subject, informant, or clinician; 2) Montreal Cognitive Assessment (MoCA) score between 19-25 and impairment in learning and memory domain; 3) essentially normal functional activities as derived from the Clinical Dementia Rating Scale (CDR) and 4) the National Institute on Aging and Alzheimer's Association (NIA-AA) criteria for MCI due to Alzheimer's disease. , Age is greater than or equal to 50 years old. Meets the National Institute on Aging and Alzheimer's Association (NIA-AA) criteria for MCI due to Alzheimer's disease.

Essentially normal functional activities as derived from the CDR. If receiving ongoing cholinesterase inhibitor therapy and/or memantine, must be on a stable dosage for at least the prior 3 months.

MoCA score between 19 and 25 at screening assessment and impairment in learning and memory domain.

Exclusion Criteria:

Cannot tolerate blood draws. Claustrophobia (fear of small or enclosed spaces), that cannot tolerate MRI scanners*.

A pace-maker or other metal implants that would preclude safe use of MRI*. DSM 5 diagnosis of alcohol or other substance use disorders within the past 12 months.

Unstable medical illness, (e.g., uncontrolled diabetes mellitus or hypertension).

Any history of stroke, seizures, MS, or Lyme disease. Any issues with ambulation, vision, or hearing which could, in the opinion of the investigator, interfere with their ability to complete assessments.

Participant does not speak English at a level necessary for the completion of the assessments.

Has not completed at least a grade eight education, as necessary for the completion of the assessments.

Currently participating in another clinical research study involving an investigational product.

History of significant agitation and/or aggression, epileptic seizures. Current neurologic disease affecting cognition other than Alzheimer's disease. Photosensitivity reactions to sunlight or visible light (polymorphous light eruption, solar urticaria, persistent light reactivity).

History of recurrent epistaxis within the last 24 weeks or currently taking major anti-coagulants (including warfarin, low molecular weight heparin) Increased skin sensitivity at the treatment site including active herpes simplex in the treatment area, history of keloid formation, or history of retinoid use in the past month.

Pregnant or lactating or planning to become pregnant. Currently undergoing infrared light therapy treatment. Any reason that, in the opinion of the investigator, might place a participant at unacceptable risk for participation in the trial.

Note: *Participants with contraindications for MRI can still enroll in the trial and participate without undergoing the MRI procedure. However, if participants do not have contraindications, undergoing the MRI is required as part of the trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Cognition | Change from pre- to post-treatment (week 0, week 9)
  Montreal Cognitive Assessment (MoCA)

SECONDARY OUTCOMES:
Blood biomarkers | Change from pre- to post-treatment (week 0, week 9)
  peripheral blood lactate and lactate/pyruvate ratio (blood draw)
Imaging biomarker | Change from pre- to post-treatment (week 0, week 9)
  Proton magnetic resonance spectroscopy (H-MRS) for brain metabolites

OTHER OUTCOMES:
Follow up cognition | Week 13 - Four weeks after the post-treatment assessments
  Montreal Cognitive Assessment (MoCA)
Follow up blood-based biomarker | Week 13 - Four weeks after the post-treatment assessments
  Blood test (lactate/pyruvate)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papi S, Allahverdipour H, Jahan A, Dianat I, Jafarabadi MA, Salimi MM. The effect of transcranial photobiomodulation on cognitive function and attentional performance of older women with mild cognitive impairment: a randomized controlled trial. Prz Menopauzalny. 2022 Sep;21(3):157-164. doi: 10.5114/pm.2022.119794. Epub 2022 Sep 28. PMID 36254133
- [Background] Cheung MC, Lee TL, Sze SL, Chan AS. Photobiomodulation improves frontal lobe cognitive functions and mental health of older adults with non-amnestic mild cognitive impairment: Case studies. Front Psychol. 2023 Jan 10;13:1095111. doi: 10.3389/fpsyg.2022.1095111. eCollection 2022. PMID 36704674
- See also: Results of the pilot study — https://www.medrxiv.org/content/10.1101/2025.08.19.25333989v1